CLINICAL TRIAL: NCT02484677
Title: Pharmacokinetics and Pharmacogenetics-based Adaptive Dosing of 5-fu (5-Fluorouracile) in Head & Neck Cancer Patient Undergoing Docetaxel, Cisplatin, 5-Fluorouracile (=TPF) Therapy
Acronym: 5-FU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-41; 2014-005536-34 (EudraCT Number); RCAPHM14_0370 (Other: APHM)
Record Dates: First submitted 2015-06-22; First posted 2015-06-30 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Patients With Head and Neck Cancer (ORL)
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Head and neck cancer patient (Experimental): Association of Docetaxel, Cisplatin, 5-Fluorouracile for pharmacokinetic evaluation
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: 5-Fluorouracile

INTERVENTIONS:
Drug: Cisplatin — Antineoplastic cytostatic. Blood sampling for pharmacokinetic evaluation
Drug: Docetaxel — Taxanes. Blood sampling for pharmacokinetic evaluation
Drug: 5-Fluorouracile — Antineoplastic and immunomodulating agents. Blood sampling for pharmacokinetic evaluation

SUMMARY:
Docetaxel, Cisplatin, 5-Fluorouracile (=TPF) is a mainstay for treating head and neck cancers, but elderly or fragile patients are often precluded because of the risk of severe toxicities associated with this protocol. DPD (Dihydro Pyrimidine Dehydrogenase) deficiency is a pharmacogenetic syndrome responsible for most of the severe/lethal toxicities showing in 5-FU (5-Fluorouracile)-treated patients, and our institute has developed a strategy for the routine determination of Dihydro Pyrimidine Dehydrogenase (DPD) status prior to starting giving the 5-FU so as to roughly adapt drug dosage according to the Dihydro Pyrimidine Dehydrogenase (DPD) status. This project aims at developing a Bayesian strategy to further individualize 5-FU dosing to reach a target exposure of area under curve (AUC). To this end, 100 patients with head and neck cancer and scheduled for a Docetaxel, Cisplatin, 5-Fluorouracile (=TPF) regimen will be included.

DETAILED DESCRIPTION:
Crop the plasma exposure of 5-FU (5-Fluorouracile) around a predefined target area under the curve 30 (AUC30) in patients with head and neck cancer treated with Docetaxel, Cisplatin, 5-Fluorouracile (=TPF) protocols and correlate adaptive Bayesian procedure to tolerability.

* Develop a population die from a group of 20 patients for which a pharmacokinetic study will be carried out
* Evaluate obtaining effective concentration of 5-FU in the context of a Docetaxel, Cisplatin, 5-Fluorouracile (=TPF) protocol adapted by the Bayesian procedure.
* Compare recommendations in terms of dosage adjustment of Bayesian approach with the recommendations of a simplified graphical approach.
* Test the measure of Dihydro Pyrimidine Dehydrogenase (DPD) activity Dihydrouracil/Uracile (UH2 / U ratio) as a co-variable adjustment of 5-Fluorouracile (5-FU) regimens in Pharmacogenomics/Pharmacokinetic (PGx / PK) model.
* Evaluate a prototype of urinary dipsticks for the early detection of toxicity from the assay as a marker of Dihydro Pyrimidine Dehydrogenase (DPD) activity.
* Assess the cost-benefit of dosage targeting, in terms of reduction resulting costs to the management of chemotherapy-induced toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and ≤ 80 years.
* Squamous cell carcinoma of the head and neck (oral cavity, oropharynx, hypopharynx, larynx, nasopharynx).
* Locally advanced stage (III, IVa or IVb).
* The patient must have received the information note and signing the informed consent, as well as being spent in multidisciplinary meeting after which treatment with TPF (Docetaxel, Cisplatin, 5-Fluorouracile) induction chemotherapy was proposed.
* Performance Status less than or equal to 2 (WHO performance index).
* The patient must be affiliated to a social security scheme and followed in one of the participating centers.
* Patients polymorphonuclear neutrophil greater than or equal to 1000 / mm3, platelets greater than or equal to 100 000 / mm3, hemoglobin greater than or equal to 8 g / dl, transaminases less than or equal to 1.5 times the normal, total bilirubin or equal 1.5 times the normal creatinine clearance in the upper or equal to 50 ml / min Modification of Diet in Renal Disease (MDRD)
* Satisfactory heart function
* Patients must be able to submit to the rhythm of visits, treatment plan, laboratory balances and other study procedures.

Exclusion Criteria:

* Patient > 80 years.
* Patients with uncontrolled infection that could compromise participation in the study.
* Patients with other serious concomitant diseases and / or uncontrolled that could compromise participation in the study.
* Patients with serum bilirubin> under limit normal and / or Alanine Transaminase (ALAT) and Aspartate Transaminase (AST) 3.5 times the under limit normal with alkaline phosphatase greater than 6 times the under limit normal.
* Cardiovascular disease or clinically significant cardiovascular disorder in the judgment of the investigator, such as, but not limited to uncontrolled hypertension, congestive heart failure The New York Heart Association (NYHA) classification> III), unstable angina, myocardial infarction in 6 months prior to treatment, uncontrolled arrhythmias, chronic liver or renal disease, severely impaired lung function.
* Disorders significant acute gastrointestinal or recent with a major symptom of diarrhea, such as Crohn's disease, malabsorption syndrome or diarrhea Common toxicity Criteria for Adverse Events (CTCAE) grade> 1 whatever aetiology.
* Performance Status and / or laboratory tests incompatible with chemotherapy using cisplatin, docetaxel and 5-fluorouracile (5-FU)
* Inability to submit to medical monitoring test for geographical reasons, family, social or psychological.
* Patients refusing to participate in biological assessments.
* Persons deprived of liberty or guardianship.
* Pregnant women or likely to be at the time of enrollment or during breastfeeding.
* Free, informed and signed not obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Determination of 5-FU (5-Fluorouracile) | 24 months
  Concentration of 5-FU in nanograms per milliliter. Circulating 5-FU will be quantified by immunoassay.
Toxicities | 24 months
  will be graded according to Common toxicity Criteria (CTC) 2.0 standards.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France